CLINICAL TRIAL: NCT07209761
Title: A Phase 3, Randomized, Open-label, Multicenter Trial to Evaluate the Efficacy, Safety, and Tolerability of 4-month and 6-month Quabodepistat-containing Regimens for Rifampicin-resistant/Multidrug-resistant Pulmonary Tuberculosis
Brief Title: A Study of Quabodepistat-containing Regimens for the Treatment of Drug-resistant Pulmonary Tuberculosis
Acronym: QUANTUM-TB
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 323-201-00013
Record Dates: First submitted 2025-08-12; First posted 2025-10-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Tuberculosis
Keywords: Pulmonary Tuberculosis; Quabodepistat; Bedaquiline; Pretomanid; Linezolid; Moxifloxacin; Fluoroquinolone-sensitive TB; Fluoroquinolone-resistant TB; Drug-resistant TB; Shortened TB treatment
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — bedaquiline; pretomanid; Moxifloxacin; Linezolid

STUDY DESIGN:
Intervention Model Description: The study has two parallel cohorts based on fluoroquinolone sensitivity status, each with an experimental arm and a control arm.
Masking Description: This is an open-label study with blinded endpoint adjudication of the primary efficacy outcome. Certain sponsor team members will be blinded to treatment assignments to minimize potential bias as much as possible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- BPaQM for Fluoroquinolone-sensitive RR/MDR-TB (Experimental): Bedaquiline 400 mg once daily for 2 weeks then 100 mg once daily for 15 weeks + Pretomanid 200 mg QD for 17 weeks + Quabodepistat 30 mg once daily for 17 weeks + Moxifloxacin 400 mg once daily for 17 weeks
  Interventions: Drug: BPaQM
- BPaLM for Fluoroquinolone-sensitive RR/MDR-TB (Active Comparator): Bedaquiline 400 mg once daily for 2 weeks then 200 mg thrice a week for 24 weeks + Pretomanid 200 mg QD for 26 weeks + Linezolid 600 mg once daily for 26 weeks + Moxifloxacin 400 mg once daily for 26 weeks
  Interventions: Drug: BPaLM
- BPaQ for Fluoroquinolone-resistant RR/MDR-TB (Experimental): Bedaquiline 400 mg once daily for 2 weeks then 100 mg once daily for 24 weeks + Pretomanid 200 mg QD for 26 weeks + Quabodepistat 30 mg once daily for 26 weeks
  Interventions: Drug: BPaQ
- BPaL for Fluoroquinolone-resistant RR/MDR-TB (Active Comparator): Bedaquiline 400 mg once daily for 2 weeks then 200 mg thrice a week for 24 weeks + Pretomanid 200 mg QD for 26 weeks + Linezolid 600 mg once daily for 26 weeks
  Interventions: Drug: BPaL

INTERVENTIONS:
Drug: BPaQM — Bedaquiline 400 mg once daily for 2 weeks then 100 mg once daily for 15 weeks + Pretomanid 200 mg QD for 17 weeks + Quabodepistat 30 mg once daily for 17 weeks + Moxifloxacin 400 mg once daily for 17 weeks
  Other Names: Bedaquiline, Pretomanid, Quabodepistat, Moxifloxacin
  Arms: BPaQM for Fluoroquinolone-sensitive RR/MDR-TB
Drug: BPaLM — Bedaquiline 400 mg once daily for 2 weeks then 200 mg thrice a week for 24 weeks + Pretomanid 200 mg QD for 26 weeks + Linezolid 600 mg once daily for 26 weeks + Moxifloxacin 400 mg once daily for 26 weeks
  Other Names: Bedaquiline, Pretomanid, Linezolid, Moxifloxacin
  Arms: BPaLM for Fluoroquinolone-sensitive RR/MDR-TB
Drug: BPaQ — Bedaquiline 400 mg once daily for 2 weeks then 100 mg once daily for 24 weeks + Pretomanid 200 mg QD for 26 weeks + Quabodepistat 30 mg once daily for 26 weeks
  Other Names: Bedaquiline, Pretomanid, Quabodepistat
  Arms: BPaQ for Fluoroquinolone-resistant RR/MDR-TB
Drug: BPaL — Bedaquiline 400 mg once daily for 2 weeks then 200 mg thrice a week for 24 weeks + Pretomanid 200 mg QD for 26 weeks + Linezolid 600 mg once daily for 26 weeks
  Other Names: Bedaquiline, Pretomanid, Linezolid
  Arms: BPaL for Fluoroquinolone-resistant RR/MDR-TB

SUMMARY:
This study aims to assess quabodepistat-based treatment regimens for RR/MDR-TB. The study will enroll adults and adolescents with rifampicin-resistant or multidrug-resistant pulmonary TB. The main goal is to see if a new drug called quabodepistat, when combined with other TB drugs, can shorten treatment duration to 4 months and be as effective and safer than current WHO endorsed treatment regimen given for 6-months. The study will compare different drug combinations in two groups of patients: those whose TB is sensitive to fluoroquinolones and those whose TB is resistant to fluoroquinolones. Participants will be randomly assigned to receive either the new treatment or the standard treatment. The study will last for 16 months for each participant and will measure how well the treatments work and how safe they are.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, open-label, multicenter trial evaluating quabodepistat-containing regimens for rifampicin-resistant/multidrug-resistant (RR/MDR) pulmonary tuberculosis (TB).

The study aims to enroll 532 participants aged 14 years and older.

The study has two main cohorts:

Fluoroquinolone-sensitive RR/MDR-TB (432 participants):

* Experimental arm: BPaQM (bedaquiline, pretomanid, quabodepistat, moxifloxacin) for 4 months
* Control arm: BPaLM (bedaquiline, pretomanid, linezolid, moxifloxacin) for 6 months

Fluoroquinolone-resistant RR/MDR-TB (100 participants):

* Experimental arm: BPaQ (bedaquiline, pretomanid, quabodepistat) for 6 months
* Control arm: BPaL (bedaquiline, pretomanid, linezolid) for 6 months

The primary efficacy endpoint is an unfavorable outcome by 12 months post-randomization.

Secondary endpoints include time to unfavorable outcome, time to sputum culture conversion, and safety/tolerability assessments. Participants will be followed for 16 months post-randomization.

The study will be conducted at approximately 40 sites in up to 12 countries.

An independent Data Monitoring Committee and Endpoint Adjudication Committee will be used in the study.

The trial aims to evaluate if quabodepistat-containing regimens can shorten treatment duration to 4 months for fluoroquinolone-sensitive RR/MDR-TB and provide a safer alternative to linezolid-containing regimens for both fluoroquinolone-sensitive and fluoroquinolone-resistant RR/MDR-TB.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥14 years
2. Body weight ≥30.0 kg
3. Able to provide written informed consent (if under 18, requires both participant assent and parent/guardian consent)
4. Documented pulmonary TB: Mtb confirmed by Xpert MTB/RIF Ultra (semi-quantitative result of 'low', 'medium', or 'high')
5. Rifampicin resistance confirmed by Xpert MTB/RIF Ultra test
6. Chest radiograph consistent with active TB disease
7. Able to provide sputum sample
8. Participants of childbearing potential must use 2 different approved birth control methods during treatment and for 12 weeks after last dose
9. Willing to have HIV test (unless previous positive result confirmed)
10. For HIV-positive participants: On stable antiretroviral regimen (dolutegravir, lamivudine/emtricitabine, tenofovir) for ≥3 months, Viral load <200 copies/mL, and CD4 count >100 cells/mL

Exclusion Criteria:

1. Known/suspected resistance to BDQ, PMD, LZD, or QBS
2. Prior treatment with BDQ, PMD, LZD, DLM, QBS, or DprE1 inhibitors for ≥1 month within past 3 months
3. Severe extrapulmonary TB
4. Abnormal laboratory values: ALT/AST >2.5×ULN, Total bilirubin >1.5×ULN, eGFR <60 mL/min/1.73m², Hemoglobin <8 g/dL, Platelets <100,000 cells/mm³, WBC <2.0×10⁹/L, ANC <1000 cells/μL, and HbA1c >9.0%
5. Pre-existing peripheral neuropathy (≥Grade 1), optic neuritis, or visual impairment
6. Co-enrollment in other therapeutic trials
7. QTcF >450 msec (males) or >470 msec (females)
8. Clinically significant cardiovascular disorders
9. Bleeding disorders
10. Conditions interfering with X-ray or sputum assessment
11. Drug allergies/hypersensitivity to study medications
12. Pregnancy or breastfeeding
13. Positive drug screen (case-by-case assessment for some substances)
14. Serious mental disorders
15. Karnofsky score <60
16. BMI <16.0 kg/m²
17. Significant comorbidities (metabolic, renal, gastrointestinal, neurological, psychiatric, endocrine, liver)
18. Pulmonary conditions other than TB (silicosis, fibrosis)
19. Active SARS-CoV-2 infection
20. Use of prohibited medications
21. Blood/plasma donation within 30 days
22. Current use of herbal remedies or traditional medicines

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-05-28 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with unfavorable outcome. | From randomization to Month 12
  Unfavorable outcome is defined as a participant experiencing at least one of the following: death, treatment failure, change in regimen, or sputum culture with growth of Mycobacterium tuberculosis at certain timepoints as follows: Failure to achieve SCC at the end of the treatment period that results in a change in anti-mycobacterial therapy or Relapse during the follow-up period (i.e., the period from end of treatment to Month 12 post-randomization.
Incidence of Grade ≥3 Treatment-Emergent Adverse Events, Serious Adverse Events, or Adverse Events Leading to Dose Reduction or Discontinuation (Safety and Tolerability). | From first dose to 2 weeks after end of treatment (Week 17 for BPaQM; Week 26 for BPaLM, BPaQ, BPaL)
  A participant experiencing at least one of the following: Grade 3 toxicity or higher treatment-emergent adverse events (TEAEs), serious TEAEs, or TEAEs leading to dose reduction or discontinuation.

SECONDARY OUTCOMES:
Time to first occurrence of any event meeting the unfavorable outcome definition. | From randomization to Month 12
  Time to the first occurrence of any event listed under the primary efficacy endpoint.
Time to sputum culture conversion. | From randomization to end of treatment (Week 17 for BPaQM; Week 26 for BPaLM, BPaQ, BPaL)
  Time from randomization to the first of two consecutive negative sputum cultures taken at least 1 week apart.
Proportion of participants with sputum culture conversion. | At Week 8 and at end of treatment (Week 17 for BPaQM; Week 26 for BPaLM, BPaQ, BPaL)
  Proportion of participants achieving sputum culture conversion, defined as two consecutive negative cultures taken at least 1 week apart.
Proportion of participants with microbiological relapse. | From end of treatment (Week 17 for BPaQM; Week 26 for BPaLM, BPaQ, BPaL) to Month 12 post-randomization
  Proportion of microbiological relapse.
Proportion of participants with adverse events of special interest (AESIs). | From first dose to 2 weeks after end of treatment (Week 17 for BPaQM; Week 26 for BPaLM, BPaQ, BPaL)
  AESIs include QTc interval prolongation, hepatotoxicity, peripheral neuropathy, optic neuritis, and hematological toxicity.
Proportion of participants with treatment-emergent adverse events (TEAEs). | From randomization through Week 68
  Proportion of participants with TEAEs, Grade 3 or higher TEAEs, and serious TEAEs.
Proportion of time during treatment spent without adverse events. | From randomization to end of treatment (Week 17 for BPaQM; Week 26 for BPaLM, BPaQ, BPaL)
  Measure of difference in AE-free time during treatment between experimental and standard of care arms.
Proportion of participants who are lost to follow-up. | From randomization through Week 68
  Measure of participant retention throughout the study period.
Proportion of participants with TB-related death. | From randomization through Week 68
  Mortality specifically related to tuberculosis.
Plasma concentrations of each analyte at scheduled visits. | From randomization through Week 17 (BPaQM and BPaQ only)
  Plasma concentrations of trial drugs in experimental arms.

OTHER OUTCOMES:
To evaluate health-related quality of life measures in the experimental and SoC arms. | From baseline to Week 52 and end of treatment (Week 17 for BPaQM; Week 26 for BPaLM, BPaQ, BPaL)
  Changes from baseline in SF-36v2 Physical and Mental Component Summary scores, SF-6D utility score, SGRQ Total score and subscores (Symptoms, Activity, and Impacts), CAAT total score and subscores (symptom burden items and daily impacts items), and descriptive summaries of PRO-CTCAE adverse event frequency, severity, and interference over time.
To estimate the difference in the proportion of unfavorable outcomes between the investigational and SoC arms at specified timepoints. | At 10 months post-treatment completion and at 16 months post-randomization
  Proportion of participants with unfavorable outcome at specified timepoints beyond the primary endpoint assessment at 12 months post-randomization to evaluate durability of treatment effect.
To estimate the difference in the proportion of microbiological relapse between the investigational and SoC arms at specified timepoints. | At 10 months post-treatment completion and at 16 months post-randomization
  Proportion of participants with microbiological relapse at specified timepoints beyond the primary endpoint assessment at 12 months post-randomization to evaluate durability of treatment effect.
To evaluate the development of resistance and cross-resistance to anti-TB drugs in all treatment arms. | From baseline through Week 68
  Proportion of participants developing drug resistance during the trial and proportion of participants developing cross-resistance between bedaquiline and quabodepistat during the trial, as determined by phenotypic drug susceptibility testing and genotyping.

CONTACTS AND LOCATIONS:
Overall Officials: Simbarashe G Takuva, MD, MSc., Study Director — Study Sponsor
Locations (33):
- China (6):
  - Capital Medical University - Beijing Chest Hospital, Beijing, Beijing Municipality
  - The Third People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Wuhan Institute of Tuberculosis Control (Wuhan Pulmonary Hospital), Wuhan, Hubei
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Shanghai Pulmonary Hospital - Pneumology, Shanghai, Shanghai Municipality
  - Public Health Clinical Center of Chengdu, Chengdu, Sichuan
- National Center for Tuberculosis and Lung Disease, Tbilisi, Georgia
- Japan Anti-Tuberculosis Association Fukujuji Hospital, Kiyose, Tokyo, Japan
- IMSP Institutul de Ftiziopneumologie Chiril Draganiuc - Phthisiopneumology, Chisinau, Chisinau City, Moldova
- Peru (3):
  - Socios en Salud Sucursal Peru, La Molina, Lima region
  - Centro de Investigación del Hospital de Emergencias de Villa el Salvador, Villa El Salvador, Lima region
  - Hospital Sergio E. Bernales, Lima
- Philippines (4):
  - Silang Specialist Medical Center, Silang, Cavite
  - Jose B. Lingad Memorial Regional Hospital, San Fernando City, Central Luzon (Region III)
  - Tropical Disease Foundation, Makati City, National Capital Region
  - Lung Center Of The Philippines, Quezon City, National Capital Region
- South Africa (13):
  - Synergy Biomed Research Institute, East London, Eastern Cape
  - Isango Lethemba TB Res Unit (CHRU) - Jose Pearson TB Hospital, Port Elizabeth, Eastern Cape
  - The Aurum Institute - Tembisa Hospital Clinical Research Centre, Johannesburg, Gauteng
  - Clinical HIV Research Unit (CHRU) - Helen Joseph Hospital, Johannesburg, Gauteng
  - Sizwe Clinical Research Site (CHRU) - Sizwe Tropical Disease Hospital,, Johannesburg, Gauteng
  - Setshaba Research Center, Pretoria, Gauteng
  - Perinatal HIV Research Unit (PHRU) - Chris Hani Baragwanath Academic Hospital, Soweto, Gauteng
  - Centre for the AIDS Programme of Research in South Africa (CAPRISA), Durban, KwaZulu-Natal
  - Klerksdorp/Tshepong Hospital Complex, Tshepong Hospital, MDR Unit, Klerksdorp, North West
  - The Aurum Institute - Rustenburg, Rustenburg, North West
  - Brooklyn Chest Hospital, Belville, Western Cape
  - UCT - Lung Infection and Immunity Unit, Cape Town, Western Cape
  - UCT Lung Institute, Cape Town, Western Cape
- South Korea (4):
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon, Incheon Metropolitan City
  - Pusan National University Hospital, Busan, Pusan-Kwangyokshi
  - Seoul National University Hospital - Pulmonology, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center - Pulmonology, Seoul, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com/

REFERENCES:
- See also: Related Info — https://trials.otsuka-us.com/